CLINICAL TRIAL: NCT05613712
Title: Chronic Inflammatory Rheumatism: Management of Comorbidities in Ambulatory Medicine
Acronym: SCORIC-A
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC22.0355
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Chronic Inflammatory Disease
Keywords: rheumatoid arthritis; spondyloarthropathy; spondylarthritis; ankylosing spondylitis; psoriatic arthritis; chronic inflammatory rheumatic diseases; comorbidities; continuity of patient care; patient compliance; adherence; non-adherence
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthropathies; Spondylarthritis; Spondylitis, Ankylosing; Arthritis, Psoriatic; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients followed by the rheumatology department of the CHU Grenoble Alpes, constituting the SCORIC group
  Interventions: Other: Patients
- Referring physician: Physicians identified as the referring physician for patients in the SCORIC group
  Interventions: Other: Referring physician

INTERVENTIONS:
Other: Patients — Description by the patients through the questionnaire of the elements limiting the good ambulatory follow-up
  Groups: Patients
Other: Referring physician — Description by the referring physicians through the questionnaire of the elements limiting the applicability of the recommendations issued by the rheumatology department of the CHU Grenoble Alpes
  Groups: Referring physician

SUMMARY:
Identification of factors limiting compliance with the recommendations established during the evaluation of the SCORIC population by the rheumatology department of the CHU Grenoble Alpes

DETAILED DESCRIPTION:
In the rheumatology department of the CHU Grenoble Alpes, Professor Baillet and other rheumatologists have set up a holistic assessment of inflammatory rheumatism (rheumatoid arthritis, spondyloarthritis and psoriatic arthritis) and associated co-morbidities in a day hospital. Based on this assessment, a hospital report is drawn up summarising the patient's treatment options, which is then sent to the patient's referring physician. They analysed the first 100 patients in the cohort and showed that 98% of patients were not up to date with their care. Their longitudinal analysis shows that patients update two thirds of the recommendations made within 12 to 18 months. Therefore, the investigators would like to assess the applicability of this screening in these patients, through a questionnaire sent to the 400 patients of the cohort and to their treating physicians.

ELIGIBILITY:
Inclusion Criteria:

* Patient cohort :
* men and women over 18 years of age
* Informed volunteers who have consented to participate in the study
* have rheumatoid arthritis, spondyloarthritis or psoriatic arthritis
* have been hospitalised in a day hospital in the rheumatology department of the Grenoble-Alpes University = SCORIC cohort of the department
* Cohort of referring physicians :
* volunteers who received informed information and consented to participate in the study
* be the referring physician of a patient of the SCORIC cohort of the rheumatology department of the South Hospital of the CHU Grenoble-Alpes

Exclusion Criteria:

* Patient cohort :
* psychiatric pathologies or history of behavioural disorders
* persons referred to in articles L1121-5 to L1121-8 of the Public Health Code
* persons under guardianship or curatorship
* not affiliated to the social security system
* minors
* Refusal to participate by the patient and/or unreturned questionnaire
* Cohort of referring physicians:
* the physician is no longer the patient's referring physician
* refusal of the doctor to participate and/or questionnaire not returned

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The SCORIC population targeted by the patient questionnaire represents all patients followed by the rheumatology department of the CHU Grenoble Alpes, having benefited from a holistic analysis of their disease and their comorbidities.
  The referring physician population will be generated from the medical records of the patients of the SCORIC cohort.
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2023-02-11 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Identification of the factors limiting compliance with the recommendations established during the evaluation of the SCORIC population by the rheumatology department of the CHU Grenoble Alpes, through questionnaires | 1 day
  Identification of the factors limiting compliance with the recommendations established during the evaluation of the SCORIC population by the rheumatology department of the CHU Grenoble Alpes

SECONDARY OUTCOMES:
Elements limiting the good ambulatory follow-up, according to the patients | 1 day
  Description by the patients through the questionnaire of the elements limiting the good ambulatory follow-up
Elements limiting the applicability of the recommendations issued by the rheumatology department of the CHU Grenoble Alpes, according to the patients | 1 day
  Description by the referring physicians through the questionnaire of the elements limiting the applicability of the recommendations issued by the rheumatology department of the CHU Grenoble Alpes

CONTACTS AND LOCATIONS:
Overall Officials: Xavier ROMAND, PHD, Principal Investigator — CHU Grenoble Alpes
Locations (1):
- CHU Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lagadou A, Gastaldi R, Vacher L, Baillet A. Gender influences adhesion to recommendations for optimal comorbidity screening and management of patients with chronic inflammatory rheumatic diseases starting a biological disease-modifying antirheumatic drug. RMD Open. 2024 Nov 11;10(4):e004364. doi: 10.1136/rmdopen-2024-004364. No abstract available. PMID 39532462